CLINICAL TRIAL: NCT03135249
Title: Sequential Natalizumab - Alemtuzumab Therapy in Patients With Relapsing Forms of Multiple Sclerosis (SUPPRESS)
Brief Title: Sequential Natalizumab - Alemtuzumab Therapy in Patients With Relapsing Forms of Multiple Sclerosis
Acronym: SUPPRESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Olaf Stuve, PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 112016-060
Record Dates: First submitted 2017-04-12; First posted 2017-05-01 (Actual); Results first posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis (MS)
MeSH Terms: conditions — Multiple Sclerosis | interventions — Alemtuzumab

STUDY DESIGN:
Intervention Model Description: To determine if treatment with alemtuzumab after natalizumab maintains or reduces the ARR in patients with RRMS. The goal of this trial is to establish a disease-free state over a 24 months period in patients who received the natalizumab-alemtuzumab sequential therapy.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Alemtuzumab treatment. (Other): Patients with relapsing-remitting multiple sclerosis previously treated with natalizumab, the following treatment arms with alemtuzumab will be implemented:
  Year One: Alemtuzumab 12 mg (1.2 ml) IV Infusion via pump over a minimum of four hours daily for five days to be given within eight hours after dilution.
  Year Two: Alemtuzumab 12 mg (1.2 ml) IV Infusion via pump over a minimum of four hours daily for three days to be given within eight hours after dilution.
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab is a humanized monoclonal therapeutic antibody that rapidly depletes cluster of differentiation 52 (CD52)+ cells.
  Other Names: Lemtrada

SUMMARY:
The purpose of this study is to determine if a sequential combination therapy of natalizumab and alemtuzumab induces peripheral tolerance and reduces the annualized relapse rate (ARR) in patients with relapsing-remitting multiple sclerosis (RRMS).

DETAILED DESCRIPTION:
To determine if treatment with alemtuzumab after natalizumab reduces the ARR in patients with RRMS. The goal of this trial is to establish a disease-free state over a 24 months period in patients who received the natalizumab-alemtuzumab sequential therapy. The target population for this study are RRMS patients nearing the end of their natalizumab treatment regimen.Participants will be recruited from four different sites. Patients who meet all inclusion/exclusion criteria will be eligible for enrollment in the study.

Alemtuzumab (Lemtrada®) will be administered at a dose of 12 mg/d by intravenous (i.v.) infusion every day for five consecutive days within 14 days of the last dose of natalizumab. After 12 months, patients will be treated with a second course of alemtuzumab 12 mg/d by intravenous (i.v.) infusion every day for three consecutive days, and participants will be followed open-label for another 12 months per standard of care. Outside the scope of this study, the intention is to follow all study participants in participating centers long-term, and to record disease activity and treatment response.

Natalizumab treatment sequesters leukocytes out of the central nervous system (CNS) into the peripheral blood. Immediate sequential alemtuzumab therapy will deplete these cells more completely than alemtuzumab monotherapy, and prevent reactivation of disease activity previously treated with natalizumab. Thus, investigators hypothesize that sequential natalizumab - alemtuzumab therapy will prevent disease activation after cessation of natalizumab, and will provide sustained disease remission in many patients.

Clinical follow up by the treating physician will occur at months 0, 3, 6, 9, 12, 18 and 24 or immediately following clinical exacerbations months. During clinical visits, comprehensive medical history data will be obtained by the treating physician. Clinical visits due to suspected exacerbations associated with CNS (central nervous system) demyelination, and associated diagnostic studies and treatments, will be covered under the medical standard of care by third party payers. A recommendation to reevaluate the patient within 3 months following the clinical event to assess for extent of recovery will be made.

Standardized MRI studies of the brain will be performed at 0, 6, 12 and 24 months. Clinical imaging studies of the brain will be performed during or immediately following the onset of a clinical exacerbation will be performed at the discretion of the site PI with scan costs covered under the medical standard of care. An end of study clinical MRI of the brain with and without contrast will be recommended to study participants at week 96 as medical standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years, inclusive.
2. Diagnosis of relapsing forms of MS using revised McDonald Criteria1.
3. Expanded Disability Status Scale (EDSS) 0 - 5.5 (note: functional system changes in cerebral (or mental) functions and in bowel and bladder functions not used in determining EDSS for protocol eligibility).
4. Has had a minimum of 12 monthly doses of continuous natalizumab therapy (300 mg/d).
5. Understands English, and gives informed consent.

Exclusion Criteria:

1. Natalizumab failure based on clinician's discretion.
2. Any prior exposure to alemtuzumab.
3. Progressive MS.
4. A diagnosis of Progressive multifocal leukoencephalopathy (PML).
5. Known hypersensitivity to alemtuzumab.
6. Initiation of new immunosuppressant treatment after the subject becomes protocol-eligible (except for corticosteroids) or enrollment in a concurrent trial with immuno-active pharmacotherapies.
7. Uncontrolled diabetes mellitus defined as HbA1c > 8% and/or requiring intensive management.
8. History of cytopenia consistent with the diagnosis of myelodysplastic syndrome.
9. Clinically significant autoimmune disease other than MS that may affect the CNS, including neuromyelitis optica (NMO), systemic lupus erythematosus (SLE), or Behcet disease.
10. Active hepatitis B or C infection or evidence of cirrhosis.
11. HIV positivity.
12. Uncontrolled viral, fungal, or bacterial infection.
13. Positive pregnancy test or inability or unwillingness to use effective means of birth control. Effective birth control is defined as:

    1. Refraining from all acts of vaginal intercourse (abstinence),
    2. Consistent use of birth control pills,
    3. Tubal sterilization or male partner who has undergone vasectomy
    4. Placement of intrauterine device
    5. Use, with every act of intercourse, of a diaphragm with contraceptive jelly and/or condoms with contraceptive foam.
14. Presence of metallic objects implanted in the body that would preclude the ability of the subject to safely have MRI exams.
15. Psychiatric illness, mental deficiency, or cognitive dysfunction making compliance with treatment or informed consent impossible.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Stuve, M.D., Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - VA North Texas Health Care System, Dallas, Texas
  - UT Southwestern Medical center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rudick RA, Stuart WH, Calabresi PA, Confavreux C, Galetta SL, Radue EW, Lublin FD, Weinstock-Guttman B, Wynn DR, Lynn F, Panzara MA, Sandrock AW; SENTINEL Investigators. Natalizumab plus interferon beta-1a for relapsing multiple sclerosis. N Engl J Med. 2006 Mar 2;354(9):911-23. doi: 10.1056/NEJMoa044396. PMID 16510745
- [Background] Polman CH, O'Connor PW, Havrdova E, Hutchinson M, Kappos L, Miller DH, Phillips JT, Lublin FD, Giovannoni G, Wajgt A, Toal M, Lynn F, Panzara MA, Sandrock AW; AFFIRM Investigators. A randomized, placebo-controlled trial of natalizumab for relapsing multiple sclerosis. N Engl J Med. 2006 Mar 2;354(9):899-910. doi: 10.1056/NEJMoa044397. PMID 16510744
- [Background] Stuve O, Marra CM, Bar-Or A, Niino M, Cravens PD, Cepok S, Frohman EM, Phillips JT, Arendt G, Jerome KR, Cook L, Grand'Maison F, Hemmer B, Monson NL, Racke MK. Altered CD4+/CD8+ T-cell ratios in cerebrospinal fluid of natalizumab-treated patients with multiple sclerosis. Arch Neurol. 2006 Oct;63(10):1383-7. doi: 10.1001/archneur.63.10.1383. PMID 17030653
- [Background] Stuve O, Marra CM, Jerome KR, Cook L, Cravens PD, Cepok S, Frohman EM, Phillips JT, Arendt G, Hemmer B, Monson NL, Racke MK. Immune surveillance in multiple sclerosis patients treated with natalizumab. Ann Neurol. 2006 May;59(5):743-7. doi: 10.1002/ana.20858. PMID 16634029
- [Background] Stuve O, Cravens PD, Frohman EM, Phillips JT, Remington GM, von Geldern G, Cepok S, Singh MP, Tervaert JW, De Baets M, MacManus D, Miller DH, Radu EW, Cameron EM, Monson NL, Zhang S, Kim R, Hemmer B, Racke MK. Immunologic, clinical, and radiologic status 14 months after cessation of natalizumab therapy. Neurology. 2009 Feb 3;72(5):396-401. doi: 10.1212/01.wnl.0000327341.89587.76. Epub 2008 Nov 5. PMID 18987352
- [Background] Kowarik MC, Pellkofer HL, Cepok S, Korn T, Kumpfel T, Buck D, Hohlfeld R, Berthele A, Hemmer B. Differential effects of fingolimod (FTY720) on immune cells in the CSF and blood of patients with MS. Neurology. 2011 Apr 5;76(14):1214-21. doi: 10.1212/WNL.0b013e3182143564. PMID 21464424
- [Background] del Pilar Martin M, Cravens PD, Winger R, Frohman EM, Racke MK, Eagar TN, Zamvil SS, Weber MS, Hemmer B, Karandikar NJ, Kleinschmidt-DeMasters BK, Stuve O. Decrease in the numbers of dendritic cells and CD4+ T cells in cerebral perivascular spaces due to natalizumab. Arch Neurol. 2008 Dec;65(12):1596-603. doi: 10.1001/archneur.65.12.noc80051. Epub 2008 Oct 13. PMID 18852339
- [Background] Bloomgren G, Richman S, Hotermans C, Subramanyam M, Goelz S, Natarajan A, Lee S, Plavina T, Scanlon JV, Sandrock A, Bozic C. Risk of natalizumab-associated progressive multifocal leukoencephalopathy. N Engl J Med. 2012 May 17;366(20):1870-80. doi: 10.1056/NEJMoa1107829. PMID 22591293
- [Background] Berger JR, Fox RJ. Reassessing the risk of natalizumab-associated PML. J Neurovirol. 2016 Aug;22(4):533-5. doi: 10.1007/s13365-016-0427-6. Epub 2016 Feb 3. PMID 26843383
- [Background] Berger JR, Fox RJ. Erratum to: Reassessing the risk of natalizumab-associated PML. J Neurovirol. 2016 Aug;22(4):536-537. doi: 10.1007/s13365-016-0431-x. No abstract available. PMID 27026534
- [Background] O'Connor PW, Goodman A, Kappos L, Lublin FD, Miller DH, Polman C, Rudick RA, Aschenbach W, Lucas N. Disease activity return during natalizumab treatment interruption in patients with multiple sclerosis. Neurology. 2011 May 31;76(22):1858-65. doi: 10.1212/WNL.0b013e31821e7c8a. Epub 2011 May 4. PMID 21543733
- [Background] Krumbholz M, Meinl I, Kumpfel T, Hohlfeld R, Meinl E. Natalizumab disproportionately increases circulating pre-B and B cells in multiple sclerosis. Neurology. 2008 Oct 21;71(17):1350-4. doi: 10.1212/01.wnl.0000327671.91357.96. PMID 18936427
- [Background] Kivisakk P, Healy BC, Viglietta V, Quintana FJ, Hootstein MA, Weiner HL, Khoury SJ. Natalizumab treatment is associated with peripheral sequestration of proinflammatory T cells. Neurology. 2009 Jun 2;72(22):1922-30. doi: 10.1212/WNL.0b013e3181a8266f. PMID 19487650
- [Background] Cohen JA, Coles AJ, Arnold DL, Confavreux C, Fox EJ, Hartung HP, Havrdova E, Selmaj KW, Weiner HL, Fisher E, Brinar VV, Giovannoni G, Stojanovic M, Ertik BI, Lake SL, Margolin DH, Panzara MA, Compston DA; CARE-MS I investigators. Alemtuzumab versus interferon beta 1a as first-line treatment for patients with relapsing-remitting multiple sclerosis: a randomised controlled phase 3 trial. Lancet. 2012 Nov 24;380(9856):1819-28. doi: 10.1016/S0140-6736(12)61769-3. Epub 2012 Nov 1. PMID 23122652
- [Background] Coles AJ, Twyman CL, Arnold DL, Cohen JA, Confavreux C, Fox EJ, Hartung HP, Havrdova E, Selmaj KW, Weiner HL, Miller T, Fisher E, Sandbrink R, Lake SL, Margolin DH, Oyuela P, Panzara MA, Compston DA; CARE-MS II investigators. Alemtuzumab for patients with relapsing multiple sclerosis after disease-modifying therapy: a randomised controlled phase 3 trial. Lancet. 2012 Nov 24;380(9856):1829-39. doi: 10.1016/S0140-6736(12)61768-1. Epub 2012 Nov 1. PMID 23122650
- [Background] Hale G, Rye PD, Warford A, Lauder I, Brito-Babapulle A. The glycosylphosphatidylinositol-anchored lymphocyte antigen CDw52 is associated with the epididymal maturation of human spermatozoa. J Reprod Immunol. 1993 Mar;23(2):189-205. doi: 10.1016/0165-0378(93)90007-5. PMID 7685389
- [Background] Xia MQ, Tone M, Packman L, Hale G, Waldmann H. Characterization of the CAMPATH-1 (CDw52) antigen: biochemical analysis and cDNA cloning reveal an unusually small peptide backbone. Eur J Immunol. 1991 Jul;21(7):1677-84. doi: 10.1002/eji.1830210714. PMID 1711975
- [Background] Rowan WC, Hale G, Tite JP, Brett SJ. Cross-linking of the CAMPATH-1 antigen (CD52) triggers activation of normal human T lymphocytes. Int Immunol. 1995 Jan;7(1):69-77. doi: 10.1093/intimm/7.1.69. PMID 7718516
- [Background] Hederer RA, Guntermann C, Miller N, Nagy P, Szollosi J, Damjanovich S, Hale G, Alexander DR. The CD45 tyrosine phosphatase regulates Campath-1H (CD52)-induced TCR-dependent signal transduction in human T cells. Int Immunol. 2000 Apr;12(4):505-16. doi: 10.1093/intimm/12.4.505. PMID 10744652
- [Background] Stauch D, Dernier A, Sarmiento Marchese E, Kunert K, Volk HD, Pratschke J, Kotsch K. Targeting of natural killer cells by rabbit antithymocyte globulin and campath-1H: similar effects independent of specificity. PLoS One. 2009;4(3):e4709. doi: 10.1371/journal.pone.0004709. Epub 2009 Mar 5. PMID 19266059
- [Background] Coles AJ, Cox A, Le Page E, Jones J, Trip SA, Deans J, Seaman S, Miller DH, Hale G, Waldmann H, Compston DA. The window of therapeutic opportunity in multiple sclerosis: evidence from monoclonal antibody therapy. J Neurol. 2006 Jan;253(1):98-108. doi: 10.1007/s00415-005-0934-5. Epub 2005 Jul 27. PMID 16044212
- [Background] CAMMS223 Trial Investigators; Coles AJ, Compston DA, Selmaj KW, Lake SL, Moran S, Margolin DH, Norris K, Tandon PK. Alemtuzumab vs. interferon beta-1a in early multiple sclerosis. N Engl J Med. 2008 Oct 23;359(17):1786-801. doi: 10.1056/NEJMoa0802670. PMID 18946064
- [Background] Hu Y, Turner MJ, Shields J, Gale MS, Hutto E, Roberts BL, Siders WM, Kaplan JM. Investigation of the mechanism of action of alemtuzumab in a human CD52 transgenic mouse model. Immunology. 2009 Oct;128(2):260-70. doi: 10.1111/j.1365-2567.2009.03115.x. PMID 19740383
- [Background] Bologna L, Gotti E, Manganini M, Rambaldi A, Intermesoli T, Introna M, Golay J. Mechanism of action of type II, glycoengineered, anti-CD20 monoclonal antibody GA101 in B-chronic lymphocytic leukemia whole blood assays in comparison with rituximab and alemtuzumab. J Immunol. 2011 Mar 15;186(6):3762-9. doi: 10.4049/jimmunol.1000303. Epub 2011 Feb 4. PMID 21296976
- [Background] Hill-Cawthorne GA, Button T, Tuohy O, Jones JL, May K, Somerfield J, Green A, Giovannoni G, Compston DA, Fahey MT, Coles AJ. Long term lymphocyte reconstitution after alemtuzumab treatment of multiple sclerosis. J Neurol Neurosurg Psychiatry. 2012 Mar;83(3):298-304. doi: 10.1136/jnnp-2011-300826. Epub 2011 Nov 5. PMID 22056965
- [Background] Cossburn MD, Harding K, Ingram G, El-Shanawany T, Heaps A, Pickersgill TP, Jolles S, Robertson NP. Clinical relevance of differential lymphocyte recovery after alemtuzumab therapy for multiple sclerosis. Neurology. 2013 Jan 1;80(1):55-61. doi: 10.1212/WNL.0b013e31827b5927. Epub 2012 Dec 12. PMID 23243077
- [Background] Coles AJ, Fox E, Vladic A, Gazda SK, Brinar V, Selmaj KW, Skoromets A, Stolyarov I, Bass A, Sullivan H, Margolin DH, Lake SL, Moran S, Palmer J, Smith MS, Compston DA. Alemtuzumab more effective than interferon beta-1a at 5-year follow-up of CAMMS223 clinical trial. Neurology. 2012 Apr 3;78(14):1069-78. doi: 10.1212/WNL.0b013e31824e8ee7. Epub 2012 Mar 21. PMID 22442431
- [Derived] Hussain RZ, Sguigna PV, Okai A, Wright C, Madinawala M, Bass AD, Cutter GR, Manouchehri N, Stuve O. The sequential natalizumab - alemtuzumab therapy in patients with relapsing forms of multiple sclerosis (SUPPRESS) trial - Part I: Rationale and objectives. J Cent Nerv Syst Dis. 2022 Aug 29;14:11795735221123911. doi: 10.1177/11795735221123911. eCollection 2022. PMID 36062026

RESULTS

PARTICIPANT FLOW:
Groups:
- Alemtuzumab Treatment.: Patients with relapsing-remitting multiple sclerosis previously treated with natalizumab, the following treatment arms with alemtuzumab will be implemented:
  Year One: Alemtuzumab 12 mg (1.2 ml) IV Infusion via pump over a minimum of four hours daily for five days to be given within eight hours after dilution.
  Year Two: Alemtuzumab 12 mg (1.2 ml) IV Infusion via pump over a minimum of four hours daily for three days to be given within eight hours after dilution.
  Alemtuzumab: Alemtuzumab is a humanized monoclonal therapeutic antibody that rapidly depletes cluster of differentiation 52 (CD52)+ cells.
Period: Overall Study
Arm/Group | Alemtuzumab Treatment.
Started | 9 (Nine patient entered the study)
Completed | 7 (Eight patient completed the study.)
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab Treatment.
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR) From the Time of Cessation of Natalizumab Treatment.
Description: The goal of this trial is to establish a disease-free state over a 24 months period in patients who received the natalizumab-alemtuzumab sequential therapy.
  ARR was the number of confirmed relapses in a year, calculated as the total number of relapses for all participants in the treatment group divided by the total participant-years of time in study.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: number of relapses in a year
Arm/Group | Alemtuzumab Treatment.
Number analyzed (Participants) | 9
number of relapses in a year | 0 [0 to 0]

2. Primary Outcome: Relapse-free Period
Description: Relapse free period, number of months until relapse, was measured only among participants who may relapse.
Time Frame: Baseline until progression up to 12 months
Population: We are intending to report the number of months until relapse and no relapses occurred. This outcome was not measured because there was no relapse.
Arm/Group | Alemtuzumab Treatment.
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of New T2 Lesions
Description: Number of new T2 lesions as measured by MRI.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Alemtuzumab Treatment.
Number analyzed (Participants) | 9
lesions | 0 (0)

4. Secondary Outcome: Number of Enlarging T2 Lesions
Description: Number of enlarging T2 lesions as measured by MRI.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Alemtuzumab Treatment.
Number analyzed (Participants) | 9
lesions | 0 (0)

5. Secondary Outcome: Number of Gadolinium (Gd)-Enhancing Lesions
Description: Number of gadolinium (Gd)-enhancing lesions as measured by MRI.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Alemtuzumab Treatment.
Number analyzed (Participants) | 9
lesions | 0 (0)

6. Other Pre Specified Outcome: Neurological Disability Outcome
Description: Neurological disability The Expanded Disability Status Scale (EDSS) will be utilized to measure the accumulation of neurological disability.
  The EDSS is a scale providing a disability score (0 to 10) based on neurological examination and information about how the patient is able to perform tasks such as long walking. Higher the score, worse the outcomes.
Time Frame: 12 months
Population: 2 patients did not complete a 12 month EDSS assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alemtuzumab Treatment.
Number analyzed (Participants) | 7
score on a scale | 3.14 (1.49)

7. Other Pre Specified Outcome: Quality of Life Outcome
Description: Quality of life (QoL) will be measured by a pre-defined, self-administered testing battery. It measures the pleasure one derives from being able to do their work well, feelings of hopelessness and difficulties in dealing with work or in doing their job effectively, and work-related, secondary exposure to extremely stressful events. Possible scores range from 0-100, with higher scores indicating a better quality of life.
Time Frame: 12 months
Population: We were not able to collect data for 2 out of 6 participants at UTSW and 3 participants at subsite were administered incorrect versions of the questionnaire which cannot be compared to the version they were supposed to and hence not analyzed for these participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alemtuzumab Treatment.
Number analyzed (Participants) | 4
score on a scale | 71.38 (21.04)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Alemtuzumab Treatment.
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT03135249/Prot_SAP_001.pdf